CLINICAL TRIAL: NCT05198258
Title: Evaluation of Implementation and Effectiveness of Neck-specific Exercise for Persistent Disability and Pain After Whiplash Injury; a Randomized Controlled Study Using a Hybrid II Design
Brief Title: Implementation and Evaluation of Neck-specific Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sormland County Council, Sweden (Other)
Collaborators: Division of Preventation,Rehabilitation av Community Science, Linköping University (Unknown); Institution of Medical Sciences, Örebro University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SormlandCCGP
Record Dates: First submitted 2022-01-04; First posted 2022-01-20 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Neck Pain; Whiplash Injuries; Neck Disorder
Keywords: Whiplash-associated disorders; Implementation Science; Neck pain; Rehabilitation; Exercise; Internet; Randomized Controlled Trial
MeSH Terms: conditions — Neck Pain; Whiplash Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study is a prospective cluster-randomized mixed-design study with hybrid II trial design.
  Twenty physiotherapy clinics in primary health care will be included.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Implementation study - experimental group (Experimental): Physiotherapists in the experimental group (group A) will receive on-line theoretical education including three hours of practical training by the project leaders. The standardized theoretical education includes three 45 minutes on-line lectures. The theoretical education will be followed by three hours practical training including clinical examination in patients with neck disability and instructions how to perform the neck-specific exercises.To facilitate the implementation process, group A will receive additional support; the physiotherapists can contact the project leader via e-mail, phone, online meetings and/or outreach visits
  Interventions: Other: Implementation strategy - experimental group
- Implementation study - control group (Active Comparator): Physiotherapists in the control group (group B) will receive the same theoretical and practical training as group A but without additional support from the research group or education after the first three theoretical on-line lectures and the three hours practical education.
  Interventions: Other: Implementation - control group

INTERVENTIONS:
Other: Implementation strategy - experimental group — On-line theoretical education and three hours of practical training by the project leaders. Contact with the project team via e-mail, phone and on-line repetition of the education for remaining of the clinical examination, neck-specific program and the progression of exercises.
  Arms: Implementation study - experimental group
Other: Implementation - control group — Physiotherapists in the control group will receive the same theoretical and practical training as the experimental group but without repetition of the education or support from the research team.
  Arms: Implementation study - control group

SUMMARY:
Persistent pain and disability in whiplash-associated disorders (WAD) grade II and III are common. Randomized controlled studies (RCTs) have shown promising result for neck-specific exercise (NSE) programmes in chronic WAD with clinically and statistically significant improvement in pain and disability. Neck-specific exercise with internet support (NSEIT) and four visits to a physiotherapist was non-inferior to NSE at a physiotherapist clinic 2 times a week in 12 weeks (24 visits). The aims of the proposed study are to evaluate an implementation strategy for NSE and NSEIT in primary health care and to evaluate the effectiveness of NSE and NSEIT in clinical practice.

DETAILED DESCRIPTION:
The study is a prospective cluster-randomized study with hybrid II trial design.

In total will 20 physiotherapy clinics in primary health care be recruited. Reg. physiotherapists working in the twenty physiotherapy clinics will be included. The clinics will be randomised to two groups with different implementation strategy: (A, intervention) three theoretical on-line lectures and the three hours' practical training with additional support; (B, control) the same education and practical training as A but with no additional support. Twenty-five patients with neck pain will be consecutively recruited from each clinic, a total of 500 patients. Outcome measurements will be conducted at baseline, 3- and 12-months.

This trial will evaluate the implementation strategy in terms of adoption of and adherence to NSEIT and NSE in clinical primary health care, also measuring diffusion of the method to other neck pain patients. In parallel, effectiveness of the exercises are evaluated.

All analyses will be conducted in collaboration with a statistician using parametric or non-parametric statistics depending on the type of data.

1. The implementation strategy will be analyzed using parametric t-test and a linear mixed model Analysis of Variance (ANOVA) or non-parametric Mann-Whitney U test and Kruskal-Wallis to evaluate differences between group A and B and change in variables over time.

   To further evaluate the implementation strategy will two focus group studies be conducted, with a purposeful sample of physiotherapists included in the cluster-randomized mixed-design study. The overall aim of these qualitative studies is to deepen the knowledge on the uptake of the new method, i.e., the NSEIT/NSE programme (adoption), the implementation in clinical practice (implementation), and how it continues to be used (maintenance).
2. The effectiveness of NSEIT and NSE will be analysed with a linear mixed model Analysis of Variance (ANOVA) or Kruskal-Wallis depending on the data.

The effect of neck-specific exercises in the present study will also be evaluated and compared to the results in our former RCT-studies.

Sample size and power regarding group differences were calculated by a statistician. Sample size calculation was based on the assumption that 15% more patients will receive neck-specific exercises in the intervention group (40% in the intervention group and 25% in the control group). The required sample size under individual randomization will be 150 patients in each arm. With ten physiotherapy clinics (clusters) in each arm (a total of 20 clusters), intra-cluster correlation of 0.02 and a cluster size of 21 patients, a total of 420 patients are recruited for 80% power and a significance level of 0.05. To ensure that enough people are in each group after dropouts, a total of 500 patients will be included, 25 patients from each cluster. The patients will be consecutively recruited.

Patients who are included in both the intervention and control groups and received neck-specific exercises will be treated as one group in terms of the effect of the intervention. The sample size calculation to evaluate effectiveness was based on a clinically relevant improvement of 7% on the Neck Disability Index (NDI), effect size 0.2 (Cohen's f) or 0.4 (Cohen's d), and correlation among repeated measures of 0.3, resulting in a total of 56 participants for 80% power and a significance level of 0.05. With an expected dropout rate of 20%, a total of 70 participating patients are needed.

The patients will be analysed as one group and the total number of patients may be more than 70 because patients will be included at each clinic. All analyses will be conducted in collaboration with a statistician using parametric or non-parametric statistics depending on the type of data. Data will be analysed according to intention to treat and supplemented with per protocol analysis.

ELIGIBILITY:
Inclusion criteria implementation

- Reg. physiotherapists working in twenty physiotherapy clinics in primary health care.

Exclusion criteria implementation

- No exclusion criterta

Inclusion criteria to evaluate the effectiveness of neck-specific exercise

* The physiotherapists will include patients ≥ 18 years with neck pain.
* Patients are required to have internet access by phone, tablet, or computer
* Be able to read and understand Swedish

Exclusion criteria:

* Physiotherapists should exclude patients with "red flags"i.e., symptoms that suggest a serious illness or spinal abnormality.
* Serious trauma to the neck and no X-ray
* Preceding neck surgery
* Osteoporosis
* Myelopathy
* History of cancer
* Unexplained weight loss
* Present fever, history of infections
* Constant and progressive non-mechanical pain
* Insidious progression of pain
* Signs of spinal cord compression (neurological examination to exclude spinal cord or cervical myelopathy such as clumsy hands, altered gait, or disturbances of sexual, bladder or sphincter function).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Implementation - Adoption of neck-specific exercise programmes | Baseline to 3 and 12 months (proportions of 500 patients with neck pain from 20 physiotherapy clinics)
  Proportion of patients with neck pain receiving neck-specific exercise
Patient Effectiveness - Neck Disability Index | Change from baseline to 3 months (after treatment) and 12 months follow-up
  Self-reported neck-specific function

SECONDARY OUTCOMES:
Implementation - The Evidence-Based Practice Attitude Scale (EBPAS) | Baseline
  Physiotherapists attitudes to implementation of evidence-based practice
Implementation - Practitioner Confidence Scale (PCS) | Change from baseline to 3 months (after treatment) and 12 months follow-up
  Self-efficacy and confidence to diagnose and treat patients with neck pain
Patient - Pain intensity (current, average last week, worst pain last week) in neck, head, and arm, and dizziness (current, average last week, worst dizziness last week) | Change from baseline to 3 months (after treatment) and 12 months follow-up
  Numeric Rating Scale (NRS); 0=no pain or dizziness, 10=worst imaginable pain or dizziness).
Patient - rating of self-perceived health | Change from baseline to 3 months (after treatment) and 12 months follow-up
  How is your current health in general? Numeric Rating Scale 0-10, 0=the worst health; 10= "the best health you can imagine
Patient - Workability | Change from baseline to 3 months (after treatment) and 12 months follow-up
  Self-reported workability measured with the Work Ability Score (WAS). The worker's self-assessment of his/her current ability to work compared to the lifetime best.WAS; (0 = currently can not work at all, 10=work ability at it's best
Patient - The patient's assessment of perceived anxiety and depression | Change from baseline to 3 months (after treatment) and 12 months follow-up
  During the last week, have you felt anxious or depressed? Numeric Rating Scale (0-10), 0=no, not at all; 10= yes, very much
Patient - Improvement or deterioration over time | Measured at 3 months and 15 months follow up
  Global Rating scale (GRS) (-5=vastly worse, 0=unchanged, 5=completely recovered)

OTHER OUTCOMES:
Background data | Baseline
  Background data from physiotherapists and patients such as age and gender
Implementation Qualitative data | After 2 and 12 months
  Two focus group studies with a purposeful sample of physiotherapists

CONTACTS AND LOCATIONS:
Overall Officials: Gunnel Peterson, Study Chair — Centre for Clinical Research Sörmland, Uppsala University, Sweden; Anneli Peolsson, Study Chair — Department of Health, Medicine and Caring Sciences, unit of Physiotherapy, Linköping University; Emma Nilsing-Strid, Study Chair — University Health Care Research Center, Faculty of Medicine and Health, Örebro University; Siw Carlfjord, Study Chair — Department of Health, Medicine and Caring Sciences, unit of Physiotherapy, Linköping University
Locations (7):
- Sweden (7):
  - Gunnel Peterson, Leksand, Dalarna County
  - Gunnel Peterson, Ljusdal, Gävleborg County
  - Gunnel Peterson, Helsingborg, Skåne County
  - Gunnel Peterson, Nyköping, Sörmland
  - Gunnel Peterson, Uppsala, Uppsala County
  - Sofia Ask, Västerås, Västmanland County
  - Emma Nilsing-Strid, Örebro

REFERENCES:
- [Derived] Peterson G, Carlfjord S, Nilsing Strid E, Ask S, Jonsson M, Peolsson A. Evaluation of implementation and effectiveness of neck-specific exercise for persistent disability and pain after whiplash injury: study protocol for a randomized controlled study using a hybrid 2 design. BMC Musculoskelet Disord. 2022 May 30;23(1):516. doi: 10.1186/s12891-022-05470-y. PMID 35637458